CLINICAL TRIAL: NCT02971462
Title: Remote Ischemic Conditioning for Reducing Stroke Risk of Symptomatic Vertebrobasilar Lesion of Atherosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ji Xunming (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming, VP,Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIC-SVAS
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Vertebrobasilar Ischemia
Keywords: stroke; Vertebrobasilar atherosclerosis; remote ischemic conditioning
MeSH Terms: conditions — Vertebrobasilar Insufficiency; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIC group (Experimental): Experimental: RIC group The upper limb ischemic conditioning is composed of five cycles of bilateral upper limb ischemia intervened by reperfusion, which is induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. This therapy started within 1 month after stroke. In addition, all participants receive a standard clinical therapy.
  Interventions: Device: ischemic conditioning
- Control group (No Intervention): The participants receive a standard clinical therapy after diagnosed ischemic stroke.

INTERVENTIONS:
Device: ischemic conditioning — In this study, the remote ischemic conditioning treatment was composed of five cycles of bilateral upper limb ischemia intervened by reperfusion, which was induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation.
  Other Names: Doctormate, IPC-906
  Arms: RIC group

SUMMARY:
The purpose of this study is to investigate whether remote ischemic conditioning(RIC) would reduce the stroke risk of patients with symptomatic vertebrobasilar lesion of atherosclerosis,then we would observe the haemodynamics and plasma biomarkers changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age from 18 to 80 years old.
* Patients having an ischemic stroke or a TIA within 30 days and with mRS score≤4 prior to randomization.
* The entry event is attributed to symptomatic atherosclerotic lesion（stenosis is greater than or equal to 50% or occlusion）in vertebrobasilar artery that is documented by magnetic resonance angiography (MRA) or computed tomographic angiography (CTA).
* Informed consent obtained.

Exclusion Criteria:

1. Thrombolytic therapy within 24 hours prior to enrollment.
2. Progressive neurological signs within 24 hours prior to enrollment.
3. Cerebral venous thrombosis/stenosis.
4. vertebrobasilar lesions due to arterial dissection, Moya Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other infection; any artery stenosis associated with cerebrospinal fluid (CSF) pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus.
5. Any of the following unequivocal cardiac source of embolism: rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with the participation.
6. Uncontrolled severe hypertension [sitting systolic blood pressure (SBP) >180 mmHg and/or sitting diastolic blood pressure (DBP) >110 mmHg after medication].
7. Patients with serious complications or abnormal laboratory parameters: aspartate transaminase (AST) and/or alanine transaminase (ALT) >3×upper limit of normal range; creatinine clearance <0.6 ml/s and/or serum creatinine >265 μmol/l (>3.0 mg/dl); platelets <100×109/L.
8. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural) within 90 days prior to enrollment.
9. Intracranial neoplasm, cerebral aneurysm or arteriovenous malformation.
10. Known retinal hemorrhage or visceral bleeding within 30 days prior to enrollment.
11. Severe hemostatic disorder or severe coagulation dysfunction.
12. Subclavian arterial stenosis≥50% or subclavian steal syndrome.
13. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform one of these procedures within 12 months after enrollment.
14. Major surgery (including open femoral, aortic, or carotid surgery, cardiac) within previous 30 days or scheduled in the 6 months after enrollment.
15. Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
16. Pregnant or breast-feeding women.
17. Unwilling to be followed up or poor compliance for treatment.
18. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.
19. Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
number of ischemic cerebrovascular events with vertebrobasilar responsibility | 0-6 months from randomization
  ischemic cerebrovascular events include ischemic stroke and transient ischemic attack

SECONDARY OUTCOMES:
number of composite outcomes events | 0-6 months from randomization
  composite outcomes events include Number of ischemic stroke ，transient ischemic attack ，cerebral hemorrhage and mortality
Number of participants with adverse events that are related to treatment | 0-6 months from randomization
number of participants with mRS 0-1 | 0-6 months from randomization
changes of hemodynamics | 0-6 months from randomization
  hemodynamics evaluation by transcranial doppler
changes of plasma biomarkers | baseline，3 and 6 months
  changes of plasma VEGF and index of thromboelastogramat at the baseline，in the first 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD. PhD, Principal Investigator — Xuanwu Hospital, Beijing